CLINICAL TRIAL: NCT05430555
Title: A Phase 1/2, First-in-Human, Open-Label, Accelerated-Titration, Two-Part Clinical Trial of TK-8001 (MAGE-A1-Directed TCR-Transduced Autologous CD8+ T-cells) in Patients With HLA-A*02:01 Genotype and Advanced-Stage/Metastatic, MAGE-A1+ Solid Tumors That Either Have No Further Approved Therapeutic Alternative(s) or Are Not Eligible for Them or Are in a Non- Curable State and Have Received a Minimum of Two Lines of Systemic Therapy
Brief Title: A Phase 1/ 2, First-in-Human, Open-Label, Accelerated-Titration, Two-Part Clinical Trial of TK-8001 in Patients With HLA-A*02:01 Genotype and Advanced-Stage/ Metastatic MAGE-A1+ Solid Tumors
Acronym: IMAG1NE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: T-knife GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TK-8001-01; 2021-004158-49 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-06-24 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced stage solid tumors; MAGE-A1; TCR-transgenic T-cells

STUDY DESIGN:
Intervention Model Description: This 2-part trial consists of Phase 1 dose-escalation and expansion and Phase 2. In escalation, 6-18 subjects will receive TK-8001 across 3 dose levels (DL). In expansion, subjects will be treated with the DL selected in escalation. Subjects without brain metastasis (Cohort 1) and subjects with brain metastases (Cohort 2) will both be included in expansion if DL3 is declared safe. Cohort 1 will include melanoma [skin or uveal], NSCLC, urothelial, breast, gastric esophageal, sarcoma, HNSCC, HCC, biliary tract, cervical, and salivary gland cancer subjects. Cohort 2 will only include melanoma [skin or uveal], NSCLC, urothelial, or breast cancer. In expansion, up to 20 additional subjects may be treated on DL3 if cleared during escalation. Up to 10 additional Cohort 2 subjects may be treated on DL3 if cleared during escalation. 33 subjects maximum may be treated on DL3 during Phase 1. If DL2 was safely completed the maximum total number of subjects to be treated on DL2 would be 12.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAGE-A1 - directed TCR transduced autologous T-cells (Experimental): Single-dose, intravenous infusion
  Interventions: Biological: Autologous CD8+ T-cells, transduced with MAGE-A1 directed TCR

INTERVENTIONS:
Biological: Autologous CD8+ T-cells, transduced with MAGE-A1 directed TCR — Single-dose intravenous infusion of MAGE-A1 directed TCR-transgenic T cells following a conditioning chemotherapy

SUMMARY:
The aim of this study is to determine the safety, tolerability and anti-tumoral activity of autologous T cells transduced with a T cell receptor specific for MAGE-A1 in eligible patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2, first-in-human, open-label, accelerated titration, two-part clinical trial of TK-8001 (MAGE-A1-directed TCR-transduced autologous CD8+ T-cells) in subjects with HLA-A*02:01 genotype and advanced stage/metastatic, MAGE-A1+ solid tumors (including but not limited to melanoma [skin or uveal], NSCLC, urothelial, breast, gastric [including gastroesophageal junction], esophageal, sarcoma, HNSCC, HCC, biliary tract, cervical, and salivary gland cancer) that either have no further approved therapeutic alternative or are not eligible for them or that are in a non-curable state as per the Investigator's assessment and have received a minimum of two lines of systemic therapy.

This two-part clinical trial will consist of a Phase 1 Part, which includes dose-escalation and expansion, and a Phase 2 Part.

In the Phase 1 Part dose-escalation, at least 6 subjects and up to 18 subjects (if DLT occurs) will receive escalating doses of TK-8001, with up to three dose levels explored. During the Phase 1 Part expansion, up to 20 additional subjects may be treated on DL3 if cleared during dose escalation to further evaluate the safety and efficacy of TK-8001 (Cohort 1).

An additional cohort of up to 10 subjects with brain metastases (Cohort 2) may also be treated on DL3 if cleared during dose-escalation. The maximum total number of subjects to be treated on DL3 during Phase 1 will be 33 subjects.

In the Phase 2 Part, up to 30 patients will receive TK-8001 to further evaluate the efficacy and safety of TK-8001 and to confirm the RP2D.

Both the Phase 1 Part and Phase 2 Part of the trial will consist of the following periods: Screening and Leukapheresis Period, Conditioning Period, TK-8001 Treatment Period, DLT Monitoring Period, Short-term Follow-up Period (Year 1), and Long-term Follow-up Period (Year 2 - 15).

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and comply with study procedures
* At least 18 years old
* Phase 1 Part dose-escalation and Phase 1 Part expansion Cohort 1 only: Presence of an advanced-stage/metastatic, solid tumor in non-curable state as per current medical knowledge, for which there is either no further approved therapeutic alternative available or the subject is not eligible for them or, for which the subject has completed a minimum of two lines of approved systemic therapy in the advanced-stage/metastatic setting.
* Phase 1 Part expansion Cohort 2 only: Presence of an advanced-stage/metastatic disease of the following indications: melanoma (skin or uveal), NSCLC, urothelial, breast cancer in non-curable state as per current medical knowledge, for which there is either no further approved therapeutic alternative available or the subject is not eligible for them or, for which the subject has completed a minimum of two lines of approved systemic therapy in the advanced-stage/metastatic setting.
* HLA-A*02:01 genotype.
* MAGE-A1+ tumor positive for MAGE-A1
* At least one measurable lesion, that can be accurately measured as per RECIST Version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Life expectancy > 3 months as assessed by the Investigator
* All toxicities related to prior therapy must have recovered to baseline or Grade ≤ 1 based on CTCAE v5.0
* Immune-related adverse events (irAEs) from previous therapies must have recovered to baseline or Grade ≤ 1

Exclusion Criteria:

* Any tumor-directed therapy within 14 days before start of conditioning therapy
* Any other MAGE-A1-targeting therapy.
* Pre-existing arrhythmia, uncontrolled angina pectoris, presently uncontrolled heart failure, or any myocardial infarction/coronary event as well as any thromboembolic event at any time < 6 months prior to screening.
* Left ventricular ejection fraction (LVEF) < 45% as measured by an echocardiogram
* History of CNS disease such as stroke, seizure, encephalitis, or multiple sclerosis (within 6 months prior to screening)
* Active allergy requiring continuous systemic medication or active infections requiring IV/PO anti-infectious therapy
* History of or clinical evidence of CNS primary tumors or metastases, unless they have been previously treated, and have been stable for at least 4 weeks prior to trial entry
* Major surgery within last 4 weeks prior to consent
* Active disease/ongoing infection with HIV, HBV, HCV, TB, syphilis, or SARS-CoV-2
* Receipt of any organ transplantation, except for transplants that do not require immunosuppression
* Any vaccine administration within 4 weeks of IP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 15 years after TK-8001 treatment (1 year short-term follow-up, 14 years long-term follow up)
  Incidence and grade of treatment-emergent adverse events (AEs) and serious adverse events (SAEs); Number and type of dose limiting toxicities (DLT)
Preliminary anti tumor activity | Up to 15 years after TK-8001 treatment, or until disease progression
  Evaluation of overall response rate (ORR), stable disease rate (SD), partial response rate (PR), and complete response (CR) rate of TK-8001 monotherapy, according to RECIST Version 1.1 and modified Response Evaluation Criteria in Solid Tumors (RECIST, V1.1) in cancer immunotherapy trials (iRECIST)

SECONDARY OUTCOMES:
End of dose escalation | 28 days after TK-8001 treatment of last patient in Phase 1
  RP2D will be determined through integrated evaluation of adverse events, serious adverse events, antitumoral activity, and evaluation of the biological and physiological effects of TK-8001 in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Behzad K Masouleh, MD, PhD, Study Director — T-knife GmbH
Locations (14):
- Belgium (4):
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc - Institut Roi Albert II, Brussels
  - Universite Libre de Bruxelles (ULB) - Institut Jules Bordet Anderlecht, Brussels
  - University Hospital Ghent, Ghent
  - Centre Hospitalier Universitaire (CHU) de Liège, Liège
- Germany (5):
  - Technische Universität Dresden (TU Dresden), Dresden, Saxony
  - Charité - Universitätsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Frankfurt, Goethe Universitat, Frankfurt
  - Klinikum der Universität München, Munich
  - Universitätsklinikum Würzburg, Würzburg
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (3):
  - Hospital Universitario Vall d´Hebrón, Barcelona
  - START Madrid-HM CIOCC, Madrid
  - Clínica Universidad de Navarra, Pamplona
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wermke M, Holderried TAW, Luke JJ, Morris VK, Alsdorf WH, Wetzko K, Andersson BS, Wistuba II, Parra ER, Hossain MB, Grund-Groschke S, Aslan K, Satelli A, Marisetty A, Satam S, Kalra M, Hukelmann J, Kursunel MA, Pozo K, Acs A, Backert L, Baumeister M, Bunk S, Wagner C, Schoor O, Mohamed AS, Mayer-Mokler A, Hilf N, Krishna D, Walter S, Tsimberidou AM, Britten CM. First-in-human dose escalation trial to evaluate the clinical safety and efficacy of an anti-MAGEA1 autologous TCR-transgenic T cell therapy in relapsed and refractory solid tumors. J Immunother Cancer. 2024 Jul 22;12(7):e008668. doi: 10.1136/jitc-2023-008668. PMID 39038917